CLINICAL TRIAL: NCT00875524
Title: Immunogenicity and Safety of ChimeriVax™ Tetravalent Dengue Vaccine in Healthy Subjects Aged 2 to 45 Years in Viet Nam
Brief Title: Study of ChimeriVax™ Tetravalent Dengue Vaccine in Healthy Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CYD22; 2014-001709-41 (EudraCT Number)
Record Dates: First submitted 2009-04-02; First posted 2009-04-03 (Estimated); Results first posted 2019-07-24 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Dengue Virus; Dengue Fever; Dengue Hemorrhagic Fever; Dengue Disease
Keywords: Dengue virus; Dengue fever; Dengue hemorrhagic fever; Dengue diseases; Dengue vaccine
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — ChimeriVax; Vi polysaccharide vaccine, typhoid

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The first and second vaccinations were administered in a blind-observer manner. The third vaccination was planned to be administered in a single-blind manner; however, due to the cancellation of the statistical analysis after the second vaccination, the third vaccination was also administered in a blind- observer manner. To ensure the blind-observer design of the 3 vaccinations, the product was prepared in a separate room whether neither the Investigator nor participant had access.
Oversight: Data Monitoring Committee: No

ARMS (2):
- CYD Dengue Vaccine Group (Experimental): Participants who received CYD dengue vaccine as first (Day 0), second (Day 0 + 6 months), and third (Day 0 + 12 months) injections. Participants were followed for 4 years after the third injection.
  Interventions: Biological: CYD dengue vaccine serotypes (1, 2, 3, 4).
- Control Vaccine Group (Sham Comparator): Participants who received the Meningococcal Polysaccharide Vaccine A + C, placebo, and Typhoid Vi polysaccharide vaccine as the first (Day 0), second (Day 0 + 6 months), and third (Day 0 + 12 months) injections, respectively. Participants were followed for 4 years after the third injection.
  Interventions: Biological: Meningococcal Polysaccharide A+C; NaCl; Typhoid Vi polysaccharide

INTERVENTIONS:
Biological: CYD dengue vaccine serotypes (1, 2, 3, 4). — 0.5 mL, Subcutaneous
  Other Names: ChimeriVax™
  Arms: CYD Dengue Vaccine Group
Biological: Meningococcal Polysaccharide A+C; NaCl; Typhoid Vi polysaccharide — Each at 0.5 mL, Subcutaneous, respectively
  Other Names: Meningococcal Polysaccharide Vaccine A+C; NaCl; Typhim Vi®
  Arms: Control Vaccine Group

SUMMARY:
This trial evaluated the use of a tetravalent vaccine against dengue.

Primary objectives:

* To describe the humoral immune response to dengue before and after each vaccination with tetravalent dengue vaccine in adults, adolescents, and children.
* To evaluate the safety of each vaccination with tetravalent dengue vaccine in the 4 age cohorts.
* To evaluate the persistence of antibodies against dengue during 5 years after the first vaccination with tetravalent dengue vaccine in the 4 age cohorts.

DETAILED DESCRIPTION:
Safety assessments included solicited reactions within 7 or 14 days after each injection, unsolicited adverse events within 28 days after each injection, and serious adverse events during the study period.

ELIGIBILITY:
Inclusion Criteria :

* Aged 2 to 45 years on the day of inclusion.
* Provision of Informed Consent/Assent Form signed by the participant (and/or by the parent or another legally acceptable representative for participants <18 years).
* Participant (and parent/guardian for participants <18 years) able to attend all scheduled visits and to comply with all trial procedures.
* For a female participant of child-bearing potential, avoid becoming pregnant (use of an effective method of contraception or abstinence) for at least 4 weeks prior to the first vaccination, until at least 4 weeks after the last vaccination.
* Participant in good health, based on medical history, physical examination and laboratory parameters.

Exclusion Criteria :

* Personal or family history of thymic pathology (thymoma), thymectomy, or myasthenia.
* For a female participant of child-bearing potential, known pregnancy or positive serum pregnancy test at Screening.
* For a female participant of child-bearing potential, known pregnancy or positive urine pregnancy test on the day of the first injection.
* Breast-feeding female participant.
* Receipt of any vaccine in the 4 weeks preceding the first trial vaccination.
* Human immunodeficiency virus, hepatitis B, or hepatitis C seropositivity in the blood sample taken at screening.
* Planned participation in another clinical trial during the first year of the study.
* Known or suspected congenital or acquired immunodeficiency, immunosuppressive therapy such as anti-cancer chemotherapy or radiation therapy within the past 6 months, or long-term systemic corticosteroids therapy.
* Known systemic hypersensitivity to any of the vaccine components or history of a life-threatening reaction to the trial vaccines or to a vaccine containing any of the same substances.
* Chronic illness at a stage that could interfere with trial conduct or completion, in the opinion of the Investigator.
* Current alcohol abuse or drug addiction that may interfere with the participant's ability to comply with trial procedures.
* Receipt of blood or blood-derived products in the past 3 months that might interfere with the assessment of immune response.
* Participant deprived of freedom by an administrative or court order, or in an emergency setting, or hospitalized without his/her consent.
* Laboratory abnormalities of at least moderate severity or clinically significant according to the Investigator in blood sample taken at screening.
* Participation in another clinical trial investigating a vaccine, drug, medical device, or a medical procedure in the 4 weeks preceding the first trial vaccination.
* Planned receipt of any vaccine in the 4 weeks following the first trial vaccination.
* Familial atopy medical history (parents, brothers, or sisters).
* Previous vaccination with meningococcal A+C or typhoid vaccines within 3 years prior to inclusion.
* History of meningococcal or typhoid infections (confirmed either clinically, serologically or microbiologically).

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2009-03 (Actual); Primary Completion 2014-08 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc
Locations (1):
- Sanofi Pasteur Investigational Site, Long Xuyen, An Giang, Vietnam

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study participants were enrolled from 18 March 2009 to 01 July 2010 at 1 clinical center in Vietnam.
Pre-assignment Details: A total of 180 participants who met all of the inclusion criteria and none of the exclusion criteria were enrolled and randomized.
Groups:
- CYD Dengue Vaccine Group: Participants who received CYD dengue vaccine as first (Day 0), second (Day 0 + 6 months), and third (Day 0 + 12 months) injection. Participants were followed for 4 years after the third injection.
Period: Overall Study
Arm/Group | CYD Dengue Vaccine Group | Control Vaccine Group
Started | 120 | 60
Received Vaccination 1 | 120 | 60
Received Vaccination 2 | 116 | 58
Received Vaccination 3 | 114 | 58
Completed | 112 | 54
Not Completed | 8 | 6
Not completed — Serious adverse event | 0 | 1
Not completed — Protocol Violation | 4 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Withdrawal by Subject | 3 | 5

BASELINE CHARACTERISTICS:
Population: The safety analysis set was defined as participants who received at least 1 dose of CYD dengue vaccine or control vaccine.
Groups:
- Control Group: Participants who received the Meningococcal Polysaccharide Vaccine A + C, placebo, and Typhoid Vi polysaccharide vaccine as the first (Day 0), second (Day 0 + 6 months), and third (Day 0 + 12 months) injections, respectively. Participants were followed for 4 years after the third injection.
- Total: Total of all reporting groups
Arm/Group | CYD Dengue Vaccine Group | Control Group | Total
Number analyzed (Participants) | 120 | 60 | 180
Age, Continuous [Mean (Standard Deviation); unit: Years] | 10.9 (8.6) | 11.8 (9.6) | 11.2 (8.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 25 | 87
  Male | 58 | 35 | 93

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Each Serotype of the Parental Dengue Virus Strain Before and Following Injection (Inj.) With CYD Dengue Tetravalent Vaccine
Description: Geometric mean titers against each serotype of the parental dengue virus strains were assessed using the dengue Plaque Reduction Neutralization Test (PRNT).
Time Frame: Pre-Inj. 1, 2, and 3 and 28 days Post-Inj. 1, 2, and 3
Population: Analysis was performed on Per-protocol analysis (PPA) set which included participants who received at least 1 dose of the study vaccine and had no protocol deviations, randomization error, blood sample not taken within the period and forbidden treatments. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dil)
Arm/Group | CYD Dengue Vaccine Group | Control Vaccine Group
Number analyzed (Participants) | 119 | 60
Titers (1/dil)
  Dengue Parental Serotype 1; Pre-Inj. 1 | 32.7 [21.6 to 49.5] | 19.6 [12 to 31.8]
  Dengue Parental Serotype 1; Post-Inj. 1 | 70.9 [44.3 to 113] | 18.8 [11.4 to 30.8]
  Dengue Parental Serotype 1; Pre-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 1; Pre-Inj. 2 | 52.2 [33.3 to 81.6] | 19.8 [11.4 to 34.3]
  Dengue Parental Serotype 1; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 1; Post-Inj. 2 | 100 [65.1 to 155] | 20.6 [11.8 to 36.0]
  Dengue Parental Serotype 1; Pre-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 1; Pre-Inj. 3 | 70.9 [45.5 to 110] | 24.6 [13.7 to 44.0]
  Dengue Parental Serotype 1; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 1; Post-Inj. 3 | 129 [90.5 to 183] | 25.3 [13.7 to 46.8]
  Dengue Parental Serotype 2; Pre-Inj. 1 | 33.1 [22.5 to 48.7] | 27.2 [15.3 to 48.1]
  Dengue Parental Serotype 2; Post-Inj. 1: number analyzed (Participants) | 119 | 59
  Dengue Parental Serotype 2; Post-Inj. 1 | 92.3 [58.5 to 145] | 25.0 [13.8 to 45.4]
  Dengue Parental Serotype 2; Pre-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 2; Pre-Inj. 2 | 74.8 [47.7 to 117] | 29.5 [16.0 to 54.4]
  Dengue Parental Serotype 2; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 2; Post-Inj. 2 | 195 [139 to 274] | 29.3 [16.0 to 53.8]
  Dengue Parental Serotype 2; Pre-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 2; Pre-Inj. 3 | 111 [74.4 to 165] | 32.3 [17.4 to 59.8]
  Dengue Parental Serotype 2; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 2; Post-Inj. 3 | 216 [163 to 286] | 30.4 [16.7 to 55.1]
  Dengue Parental Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 119 | 59
  Dengue Parental Serotype 3; Pre-Inj. 1 | 31.9 [23.3 to 43.8] | 20.5 [13.2 to 31.9]
  Dengue Parental Serotype 3; Post-Inj. 1: number analyzed (Participants) | 119 | 59
  Dengue Parental Serotype 3; Post-Inj. 1 | 95.6 [67.2 to 136] | 18.4 [12.0 to 28.2]
  Dengue Parental Serotype 3; Pre-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 3; Pre-Inj. 2 | 60.4 [41.9 to 87.2] | 19.1 [12.1 to 30.3]
  Dengue Parental Serotype 3; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 3; Post-Inj. 2 | 152 [115 to 203] | 21.9 [14.1 to 34.0]
  Dengue Parental Serotype 3; Pre-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 3; Pre-Inj. 3 | 87.2 [62.5 to 122] | 26.8 [17.1 to 42.1]
  Dengue Parental Serotype 3; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 3; Post-Inj. 3 | 169 [134 to 214] | 25.2 [16.3 to 39.1]
  Dengue Parental Serotype 4; Pre-Inj. 1: number analyzed (Participants) | 119 | 59
  Dengue Parental Serotype 4; Pre-Inj. 1 | 17.0 [12.8 to 22.5] | 13.9 [9.28 to 20.9]
  Dengue Parental Serotype 4; Post-Inj. 1 | 104 [71.0 to 153] | 15.4 [10.2 to 23.3]
  Dengue Parental Serotype 4; Pre-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 4; Pre-Inj. 2 | 51.7 [37.0 to 72.2] | 14.1 [9.29 to 21.4]
  Dengue Parental Serotype 4; Post-Inj. 2: number analyzed (Participants) | 115 | 57
  Dengue Parental Serotype 4; Post-Inj. 2 | 120 [89.2 to 160] | 14.3 [9.44 to 21.6]
  Dengue Parental Serotype 4; Pre-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 4; Pre-Inj. 3 | 70.1 [52.2 to 94.1] | 17.1 [10.9 to 26.9]
  Dengue Parental Serotype 4; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 4; Post-Inj. 3 | 146 [115 to 184] | 17.4 [11.2 to 27.0]

2. Primary Outcome: Geometric Mean Titers (GMTs) of Antibodies Against Each Serotype of the Parental Dengue Virus Strain During the Follow-up Period
Description: GMT against each serotype of the parental dengue virus strains were assessed using the dengue PRNT.
Time Frame: Year 1, Year 2, Year 3 and Year 4 after the Third Injection
Population: Analysis was performed on Full analysis set which included all the participants present at first vaccination (V01) and received at least one dose of vaccine. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers (1/dil)
Arm/Group | CYD Dengue Vaccine Group | Control Vaccine Group
Number analyzed (Participants) | 120 | 60
Titers (1/dil)
  Dengue Parental Serotype 1: Year 1: number analyzed (Participants) | 113 | 57
  Dengue Parental Serotype 1: Year 1 | 103 [69.0 to 152] | 28.4 [15.5 to 52.3]
  Dengue Parental Serotype 1: Year 2: number analyzed (Participants) | 112 | 57
  Dengue Parental Serotype 1: Year 2 | 72.9 [48.9 to 109] | 25.7 [14.0 to 47.3]
  Dengue Parental Serotype 1: Year 3: number analyzed (Participants) | 112 | 55
  Dengue Parental Serotype 1: Year 3 | 56.0 [35.9 to 87.4] | 29.7 [15.3 to 57.7]
  Dengue Parental Serotype 1: Year 4: number analyzed (Participants) | 112 | 54
  Dengue Parental Serotype 1: Year 4 | 52.6 [34.0 to 81.2] | 30.5 [15.8 to 58.6]
  Dengue Parental Serotype 2: Year 1: number analyzed (Participants) | 113 | 57
  Dengue Parental Serotype 2: Year 1 | 133 [91.7 to 192] | 36.9 [19.6 to 69.4]
  Dengue Parental Serotype 2: Year 2: number analyzed (Participants) | 112 | 57
  Dengue Parental Serotype 2: Year 2 | 118 [79.3 to 176] | 42.6 [22.1 to 82.0]
  Dengue Parental Serotype 2: Year 3: number analyzed (Participants) | 112 | 55
  Dengue Parental Serotype 2: Year 3 | 78.1 [52.6 to 116] | 45.2 [23.7 to 86.1]
  Dengue Parental Serotype 2: Year 4: number analyzed (Participants) | 112 | 54
  Dengue Parental Serotype 2: Year 4 | 73.7 [49.3 to 110] | 50.7 [26.5 to 97.1]
  Dengue Parental Serotype 3: Year 1: number analyzed (Participants) | 113 | 57
  Dengue Parental Serotype 3: Year 1 | 145 [104 to 202] | 31.8 [18.2 to 55.5]
  Dengue Parental Serotype 3: Year 2: number analyzed (Participants) | 112 | 57
  Dengue Parental Serotype 3: Year 2 | 88.2 [64.6 to 120] | 26.1 [15.7 to 43.7]
  Dengue Parental Serotype 3: Year 3: number analyzed (Participants) | 112 | 55
  Dengue Parental Serotype 3: Year 3 | 66.6 [47.8 to 92.9] | 24.4 [14.9 to 40.1]
  Dengue Parental Serotype 3: Year 4: number analyzed (Participants) | 112 | 54
  Dengue Parental Serotype 3: Year 4 | 42.7 [31.2 to 58.5] | 19.7 [12.5 to 31.1]
  Dengue Parental Serotype 4: Year 1: number analyzed (Participants) | 113 | 57
  Dengue Parental Serotype 4: Year 1 | 87.5 [67.2 to 114] | 19.0 [12.0 to 30.3]
  Dengue Parental Serotype 4: Year 2: number analyzed (Participants) | 112 | 57
  Dengue Parental Serotype 4: Year 2 | 56.9 [44.9 to 72.1] | 17.5 [10.9 to 27.9]
  Dengue Parental Serotype 4: Year 3: number analyzed (Participants) | 112 | 55
  Dengue Parental Serotype 4: Year 3 | 47.3 [36.9 to 60.5] | 21.7 [13.3 to 35.4]
  Dengue Parental Serotype 4: Year 4: number analyzed (Participants) | 112 | 54
  Dengue Parental Serotype 4: Year 4 | 30.2 [23.9 to 38.3] | 18.2 [11.5 to 28.8]

3. Primary Outcome: Percentage of Participants With Antibody Titers >= 10 (1/Dil) Against Each Serotypes of the Parental Dengue Virus Strains Following Inj. With CYD Dengue Tetravalent Vaccine
Description: Antibody titer levels against each serotype of the parental dengue virus strains were assessed using the PRNT.
Time Frame: Pre-Inj. 1, 2, and 3 and 28 days Post-Inj. 1, 2, and 3
Population: Analysis was performed on PPA set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Vaccine Group
Number analyzed (Participants) | 119 | 60
Percentage of participants
  Dengue Parental Serotype 1; Pre-Inj. 1 | 50.4 | 43.3
  Dengue Parental Serotype 1; Post-Inj. 1 | 62.2 | 41.7
  Dengue Parental Serotype 1; Pre-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 1; Pre-Inj. 2 | 58.3 | 39.7
  Dengue Parental Serotype 1; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 1; Post-Inj. 2 | 79.1 | 41.4
  Dengue Parental Serotype 1; Pre-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 1; Pre-Inj. 3 | 68.4 | 46.6
  Dengue Parental Serotype 1; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 1; Post-Inj. 3 | 93.0 | 41.4
  Dengue Parental Serotype 2; Pre-Inj. 1 | 49.6 | 41.7
  Dengue Parental Serotype 2; Post-Inj. 1: number analyzed (Participants) | 119 | 59
  Dengue Parental Serotype 2; Post-Inj. 1 | 66.4 | 35.6
  Dengue Parental Serotype 2; Pre-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 2; Pre-Inj. 2 | 63.5 | 39.7
  Dengue Parental Serotype 2; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 2; Post-Inj. 2 | 93.9 | 41.4
  Dengue Parental Serotype 2; Pre-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 2; Pre-Inj. 3 | 80.7 | 43.1
  Dengue Parental Serotype 2; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 2; Post-Inj. 3 | 99.1 | 43.1
  Dengue Parental Serotype 3; Pre-Inj. 1: number analyzed (Participants) | 119 | 59
  Dengue Parental Serotype 3; Pre-Inj. 1 | 63.0 | 52.5
  Dengue Parental Serotype 3; Post-Inj. 1: number analyzed (Participants) | 119 | 59
  Dengue Parental Serotype 3; Post-Inj. 1 | 84.9 | 47.5
  Dengue Parental Serotype 3; Pre-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 3; Pre-Inj. 2 | 73.0 | 46.6
  Dengue Parental Serotype 3; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 3; Post-Inj. 2 | 94.8 | 53.4
  Dengue Parental Serotype 3; Pre-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 3; Pre-Inj. 3 | 85.1 | 62.1
  Dengue Parental Serotype 3; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 3; Post-Inj. 3 | 99.1 | 58.6
  Dengue Parental Serotype 4; Pre-Inj. 1: number analyzed (Participants) | 119 | 59
  Dengue Parental Serotype 4; Pre-Inj. 1 | 44.5 | 37.3
  Dengue Parental Serotype 4; Post-Inj. 1 | 77.3 | 41.7
  Dengue Parental Serotype 4; Pre-Inj. 2: number analyzed (Participants) | 115 | 58
  Dengue Parental Serotype 4; Pre-Inj. 2 | 73.0 | 39.7
  Dengue Parental Serotype 4; Post-Inj. 2: number analyzed (Participants) | 115 | 57
  Dengue Parental Serotype 4; Post-Inj. 2 | 89.6 | 40.4
  Dengue Parental Serotype 4; Pre-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 4; Pre-Inj. 3 | 84.2 | 43.1
  Dengue Parental Serotype 4; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Dengue Parental Serotype 4; Post-Inj. 3 | 95.6 | 43.1

4. Primary Outcome: Percentage of Participants With Antibody Titers >= 10 (1/Dil) Against Each Serotypes of the Parental Dengue Virus Strains Following Inj. With CYD Dengue Tetravalent Vaccine During the Follow-up Period
Description: Antibody titer levels against each serotype of the parental dengue virus strains were assessed using the PRNT.
Time Frame: Year 1, Year 2, Year 3 and Year 4 after the Third Injection
Population: Analysis was performed on Full analysis set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Vaccine Group
Number analyzed (Participants) | 120 | 60
Percentage of participants
  Dengue Parental Serotype 1: Year 1: number analyzed (Participants) | 113 | 57
  Dengue Parental Serotype 1: Year 1 | 78.8 | 43.9
  Dengue Parental Serotype 1: Year 2: number analyzed (Participants) | 112 | 57
  Dengue Parental Serotype 1: Year 2 | 74.1 | 38.6
  Dengue Parental Serotype 1: Year 3: number analyzed (Participants) | 112 | 55
  Dengue Parental Serotype 1: Year 3 | 59.8 | 40.0
  Dengue Parental Serotype 1: Year 4: number analyzed (Participants) | 112 | 54
  Dengue Parental Serotype 1: Year 4 | 61.6 | 40.7
  Dengue Parental Serotype 2: Year 1: number analyzed (Participants) | 113 | 57
  Dengue Parental Serotype 2: Year 1 | 86.7 | 47.4
  Dengue Parental Serotype 2: Year 2: number analyzed (Participants) | 112 | 57
  Dengue Parental Serotype 2: Year 2 | 82.1 | 49.1
  Dengue Parental Serotype 2: Year 3: number analyzed (Participants) | 112 | 55
  Dengue Parental Serotype 2: Year 3 | 70.5 | 50.9
  Dengue Parental Serotype 2: Year 4: number analyzed (Participants) | 112 | 54
  Dengue Parental Serotype 2: Year 4 | 68.8 | 53.7
  Dengue Parental Serotype 3: Year 1: number analyzed (Participants) | 113 | 57
  Dengue Parental Serotype 3: Year 1 | 92.9 | 54.4
  Dengue Parental Serotype 3: Year 2: number analyzed (Participants) | 112 | 57
  Dengue Parental Serotype 3: Year 2 | 86.6 | 54.4
  Dengue Parental Serotype 3: Year 3: number analyzed (Participants) | 112 | 55
  Dengue Parental Serotype 3: Year 3 | 75.0 | 54.5
  Dengue Parental Serotype 3: Year 4: number analyzed (Participants) | 112 | 54
  Dengue Parental Serotype 3: Year 4 | 70.5 | 44.4
  Dengue Parental Serotype 4: Year 1: number analyzed (Participants) | 113 | 57
  Dengue Parental Serotype 4: Year 1 | 88.5 | 47.4
  Dengue Parental Serotype 4: Year 2: number analyzed (Participants) | 112 | 57
  Dengue Parental Serotype 4: Year 2 | 90.2 | 40.4
  Dengue Parental Serotype 4: Year 3: number analyzed (Participants) | 112 | 55
  Dengue Parental Serotype 4: Year 3 | 87.5 | 47.3
  Dengue Parental Serotype 4: Year 4: number analyzed (Participants) | 112 | 54
  Dengue Parental Serotype 4: Year 4 | 76.8 | 42.6

5. Primary Outcome: Percentage of Participants With Solicited Inj. Site Reactions Following Any and Each Inj. With CYD Dengue Tetravalent Vaccine
Description: Solicited Inj. site reactions: Pain, Erythema, and Swelling. Pain:- Grade 1: easily tolerated, Grade 2: sufficiently discomforting to interfere with normal behavior or activities, Grade 3: Incapacitating, unable to perform usual activities. Erythema and Swelling:- Grade 1: <2.5 cm, Grade 2: >=2.5 to <5 cm, Grade 3: >= 5 cm.
Time Frame: 7 days post-each injection
Population: Analysis was performed on Safety analysis set. Here, 'number analyzed' = participants with available data for each specified category.
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Vaccine Group
Number analyzed (Participants) | 120 | 60
Percentage of participants
  Inj. site Pain; Post-Any Inj. | 28.3 | 80
  Grade 3 Inj. site Pain; Post-Any Inj. | 0.0 | 0.0
  Inj. site Erythema; Post-Any Inj. | 6.7 | 21.7
  Grade 3 Inj. site Erythema; Post-Any Inj. | 0.0 | 1.7
  Inj. site Swelling; Post-Any Inj.: number analyzed (Participants) | 119 | 60
  Inj. site Swelling; Post-Any Inj. | 4.2 | 15.0
  Grade 3 Inj. site Swelling; Post-Any Inj.: number analyzed (Participants) | 119 | 60
  Grade 3 Inj. site Swelling; Post-Any Inj. | 0.0 | 1.7
  Inj. site Pain; Post-Inj. 1 | 15.8 | 73.3
  Grade 3 Inj. site Pain; Post-Inj. 1 | 0.0 | 0.0
  Inj. site Erythema; Post-Inj. 1 | 4.2 | 16.7
  Grade 3 Inj. site Erythema; Post-Inj. 1 | 0.0 | 1.7
  Inj. site Swelling; Post-Inj. 1: number analyzed (Participants) | 119 | 60
  Inj. site Swelling; Post-Inj. 1 | 1.7 | 6.7
  Grade 3 Inj. site Swelling; Post-Inj. 1: number analyzed (Participants) | 119 | 60
  Grade 3 Inj. site Swelling; Post-Inj. 1 | 0.0 | 1.7
  Inj. site Pain; Post-Inj. 2: number analyzed (Participants) | 116 | 58
  Inj. site Pain; Post-Inj. 2 | 15.5 | 15.5
  Grade 3 Inj. site Pain; Post-Inj. 2: number analyzed (Participants) | 116 | 58
  Grade 3 Inj. site Pain; Post-Inj. 2 | 0.0 | 0.0
  Inj. site Erythema; Post-Inj. 2: number analyzed (Participants) | 116 | 58
  Inj. site Erythema; Post-Inj. 2 | 4.3 | 5.2
  Grade 3 Inj. site Erythema; Post-Inj. 2: number analyzed (Participants) | 116 | 58
  Grade 3 Inj. site Erythema; Post-Inj. 2 | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 2: number analyzed (Participants) | 116 | 58
  Inj. site Swelling; Post-Inj. 2 | 2.6 | 3.4
  Grade 3 Inj. site Swelling; Post-Inj. 2: number analyzed (Participants) | 116 | 58
  Grade 3 Inj. site Swelling; Post-Inj. 2 | 0.0 | 0.0
  Inj. site Pain; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Inj. site Pain; Post-Inj. 3 | 11.4 | 41.4
  Grade 3 Inj. site Pain; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Grade 3 Inj. site Pain; Post-Inj. 3 | 0.0 | 0.0
  Inj. site Erythema; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Inj. site Erythema; Post-Inj. 3 | 2.6 | 5.2
  Grade 3 Inj. site Erythema; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Grade 3 Inj. site Erythema; Post-Inj. 3 | 0.0 | 0.0
  Inj. site Swelling; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Inj. site Swelling; Post-Inj. 3 | 0.0 | 6.9
  Grade 3 Inj. site Swelling; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Grade 3 Inj. site Swelling; Post-Inj. 3 | 0.0 | 0.0

6. Primary Outcome: Percentage of Participants With Solicited Systemic Reactions Following Any and Each Inj. With CYD Dengue Tetravalent Vaccine
Description: Solicited systemic reactions: Fever, Headache, Malaise, Myalgia, and Asthenia. Fever:- Grade 1: >=37.5 degree Celsius (°C) to <=38.0°C, Grade 2: >38.0°C to <=39.0°C, Grade 3: >39.0°C. Headache, malaise, myalgia and asthenia: Grade 1: noticeable but does not interfere with daily activities, Grade 2: interferes with daily activities, Grade 3: prevents daily activities.
Time Frame: 14 days post-each injection
Population: as for outcome 5
Measure: Number; unit: Percentage of participants
Arm/Group | CYD Dengue Vaccine Group | Control Vaccine Group
Number analyzed (Participants) | 120 | 60
Percentage of participants
  Fever; Post-Any Inj. | 27.5 | 26.7
  Grade 3 Fever; Post-Any Inj. | 0.8 | 3.3
  Headache; Post-Any Inj.: number analyzed (Participants) | 119 | 60
  Headache; Post-Any Inj. | 35.3 | 30.0
  Grade 3 Headache; Post-Any Inj.: number analyzed (Participants) | 119 | 60
  Grade 3 Headache; Post-Any Inj. | 0.8 | 0.0
  Malaise; Post-Any Inj.: number analyzed (Participants) | 119 | 60
  Malaise; Post-Any Inj. | 29.4 | 23.3
  Grade 3 Malaise; Post-Any Inj.: number analyzed (Participants) | 119 | 60
  Grade 3 Malaise; Post-Any Inj. | 0.0 | 0.0
  Myalgia; Post-Any Inj.: number analyzed (Participants) | 119 | 60
  Myalgia; Post-Any Inj. | 20.2 | 23.3
  Grade 3 Myalgia; Post-Any Inj.: number analyzed (Participants) | 119 | 60
  Grade 3 Myalgia; Post-Any Inj. | 0.0 | 0.0
  Asthenia; Post-Any Inj.: number analyzed (Participants) | 119 | 60
  Asthenia; Post-Any Inj. | 13.4 | 5.0
  Grade 3 Asthenia; Post-Any Inj.: number analyzed (Participants) | 119 | 60
  Grade 3 Asthenia; Post-Any Inj. | 1.7 | 0.0
  Fever; Post-Inj. 1 | 19.2 | 15.0
  Grade 3 Fever; Post-Inj. 1 | 0.8 | 3.3
  Headache; Post-Inj. 1: number analyzed (Participants) | 119 | 60
  Headache; Post-Inj. 1 | 29.4 | 28.3
  Grade 3 Headache; Post-Inj. 1: number analyzed (Participants) | 119 | 60
  Grade 3 Headache; Post-Inj. 1 | 0.8 | 0.0
  Malaise; Post-Inj. 1: number analyzed (Participants) | 119 | 60
  Malaise; Post-Inj. 1 | 21.8 | 16.7
  Grade 3 Malaise; Post-Inj. 1: number analyzed (Participants) | 119 | 60
  Grade 3 Malaise; Post-Inj. 1 | 0.0 | 0.0
  Myalgia; Post-Inj. 1: number analyzed (Participants) | 119 | 60
  Myalgia; Post-Inj. 1 | 15.1 | 20.0
  Grade 3 Myalgia; Post-Inj. 1: number analyzed (Participants) | 119 | 60
  Grade 3 Myalgia; Post-Inj. 1 | 0.0 | 0.0
  Asthenia; Post-Inj. 1: number analyzed (Participants) | 119 | 60
  Asthenia; Post-Inj. 1 | 8.4 | 0.0
  Grade 3 Asthenia; Post-Inj. 1: number analyzed (Participants) | 119 | 60
  Grade 3 Asthenia; Post-Inj. 1 | 0.8 | 0.0
  Fever; Post-Inj. 2: number analyzed (Participants) | 116 | 58
  Fever; Post-Inj. 2 | 12.1 | 6.9
  Grade 3 Fever; Post-Inj. 2: number analyzed (Participants) | 116 | 58
  Grade 3 Fever; Post-Inj. 2 | 0.0 | 0.0
  Headache; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Headache; Post-Inj. 2 | 15.7 | 8.6
  Grade 3 Headache; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Grade 3 Headache; Post-Inj. 2 | 0.0 | 0.0
  Malaise; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Malaise; Post-Inj. 2 | 13.0 | 8.6
  Grade 3 Malaise; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Grade 3 Malaise; Post-Inj. 2 | 0.0 | 0.0
  Myalgia; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Myalgia; Post-Inj. 2 | 9.6 | 5.2
  Grade 3 Myalgia; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Grade 3 Myalgia; Post-Inj. 2 | 0.0 | 0.0
  Asthenia; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Asthenia; Post-Inj. 2 | 6.1 | 1.7
  Grade 3 Asthenia; Post-Inj. 2: number analyzed (Participants) | 115 | 58
  Grade 3 Asthenia; Post-Inj. 2 | 0.9 | 0.0
  Fever; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Fever; Post-Inj. 3 | 3.5 | 8.6
  Grade 3 Fever; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Grade 3 Fever; Post-Inj. 3 | 0.0 | 0.0
  Headache; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Headache; Post-Inj. 3 | 8.8 | 10.3
  Grade 3 Headache; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Grade 3 Headache; Post-Inj. 3 | 0.0 | 0.0
  Malaise; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Malaise; Post-Inj. 3 | 5.3 | 8.6
  Grade 3 Malaise; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Grade 3 Malaise; Post-Inj. 3 | 0.0 | 0.0
  Myalgia; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Myalgia; Post-Inj. 3 | 4.4 | 10.3
  Grade 3 Myalgia; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Grade 3 Myalgia; Post-Inj. 3 | 0.0 | 0.0
  Asthenia; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Asthenia; Post-Inj. 3 | 0.9 | 3.4
  Grade 3 Asthenia; Post-Inj. 3: number analyzed (Participants) | 114 | 58
  Grade 3 Asthenia; Post-Inj. 3 | 0.0 | 0.0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events (SAEs) data were collected throughout the study from Day 0 to Year 4, and non-serious Adverse Events were collected for 28 days after each injection.
Description: Non-related SAEs were collected from Day 0 (post-injection) up to 6 months after the last injection. Related and fatal SAEs were reported from 6 months until the end of study (up to 4 years).
Arm/Group | CYD Dengue Vaccine Group | Control Vaccine Group
All-Cause Mortality (participants affected / at risk) | 0/120 | 0/60
Serious Adverse Events (participants affected / at risk) | 3/120 | 3/60
Other Adverse Events (participants affected / at risk) | 42/120 | 48/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=120) | Control Vaccine Group (N=60)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dengue fever (Infections and infestations) | 1 (1) | 3 (3)
Pharyngitis (Infections and infestations) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | CYD Dengue Vaccine Group (N=120) | Control Vaccine Group (N=60)
Headache; Post-Any Injection (Nervous system disorders) | 42/119 (63) | 18 (28)
Injection site Pain; Post-Any (General disorders) | 34 (50) | 48 (77)
Injection site Erythema; Post-Any (General disorders) | 8 (13) | 13 (16)
Injection site Swelling; Post-Any (General disorders) | 5/119 (5) | 9 (10)
Fever; Post-Any Injection (General disorders) | 33 (41) | 16 (18)
Malaise; Post-Any Injection (General disorders) | 35/119 (47) | 14 (20)
Asthenia; Post-Any Injection (General disorders) | 16/119 (18) | 3 (3)
Myalgia; Post-Any Injection (Musculoskeletal and connective tissue disorders) | 24/119 (34) | 14 (21)
Nasopharyngitis (Infections and infestations) | 0 (0) | 3 (3)
Pharyngitis (Infections and infestations) | 9 (9) | 7 (7)

LIMITATIONS AND CAVEATS:
None reported.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.